CLINICAL TRIAL: NCT00832949
Title: Exploring the Learning Needs of Individuals With Inflammatory Arthritis From the Perspectives of Patients, Family Members and Friends, and Health Care Providers: Patient Perspectives (One-on-one Interviews)
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Arthritis Network (Network)
Responsible Party: Mary J Bell, Sunnybrook Health Sciences Centre
Other Study IDs: DOCH2 448-2008
Record Dates: First submitted 2009-01-26; First posted 2009-01-30 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2011-01

CONDITIONS: Arthritis
Keywords: Mixed methods research (qualitative and quantitative); Peer support; Early inflammatory arthritis; Self-management; Patient education
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
Inflammatory arthritis (IA) is a major cause of long-term disability. Due to specialist shortages, failure of primary care providers and individuals to recognize the disease, and lack of awareness of the importance of early intervention, delays to rheumatologic care are common. Peer support models have been used for various health issues and may be one method to assist individuals with early IA to manage their disease and cope with stress. Qualitative research methods (one-on-one interviews) will seek out feedback on a peer support approach and explore the learning needs (informational needs, educational preferences) and opinions about emotional and appraisal support of individuals living with IA, from the perspectives of patients. The data will be analyzed and expressed themes (articulated needs and understandings of interviewee context) will guide the future development of a peer support intervention.

DETAILED DESCRIPTION:
Research Protocol

Exploring the Learning Needs of Individuals with Inflammatory Arthritis from the Perspectives of Patients, Family Members and Friends, and Health Care Providers Patient Perspectives (One-on-One Interviews) Abstract The purpose of this study is to determine the learning needs of individuals living with inflammatory arthritis from the perspective of newly diagnosed patients. Specifically, we will be looking at how culture influences the learning needs of arthritis patients. This is part of a larger study which will examine the perspectives of patients, their family members and friends, and health care providers in an effort to develop peer support methods that will improve care for individuals with inflammatory arthritis. A qualitative methodology will be utilized including semi-structured interviews. Adults with inflammatory arthritis, from different cultural groups, will be recruited to participate in the study as key informants. They will provide insight into culturally specific learning needs of different groups, which will be used to design peer support programs to better meet the needs of our increasingly diverse population.

I. Rationale Arthritis and related diseases are a group of disorders that affect joints, ligaments, bones, tendons and other parts of the musculoskeletal system (1). In Ontario, arthritis is a leading cause of pain, physical disability and use of health care services (2, 3). Although the disease is not usually life threatening, symptoms of pain, swelling and stiffness can significantly reduce quality of life and contribute to long-term disability (4). Since arthritis is a chronic disease, it must be managed throughout a patient's lifetime, with appropriate treatments for each stage of the disease. Management is usually focused on symptom control, prevention of pain and disability and improving quality of life (1).

Comprehensive care of patients with arthritis and their families includes primary care (consisting of medications, specialist and hospital care), community support services, and health education and prevention. Patient education interventions to help individuals self-manage their disease have been shown to be 20-30% as effective as pharmaceutical therapies at pain reduction and 40% as effective in reducing disability from arthritis (5). This results in decreased number of physician consultations, thereby reducing the cost of treatment for arthritis (6). Peer support is one form of patient education that may have application for arthritis patients. Components of peer support include emotional support, appraisal support and information support from a peer who shares common characteristics with the individual or group of interest (7). It is hoped that this support will help individuals with arthritis improve self-management of their disease, by helping them cope with their arthritis and become more active in managing their disease (4).

For these programs to be effective, the peer population needs to be as similar as possible to the patient population (7).Therefore, it is important to assess the needs of individuals of various cultural backgrounds in order to design programs that best address culture-specific needs and issues in the treatment of chronic disease such as arthritis. Existing recruitment strategies are often biased towards those from white, middle-class backgrounds, but more marginalized groups, including immigrants, may have the most to gain from peer support programs (8). Additionally, it has been shown that the incidence, severity and processes of care, as well as outcomes, differ among racial or ethnic groups although the reasons for this are largely unknown (9). With the diversity of the Canadian population and aging of immigrants, these are aspects that are increasingly relevant. Therefore, the design of tailored programs for different communities is important to be able to successfully implement peer support programs.

Currently, immigrants make up a significant proportion of Ontario's population. Assessing their needs after diagnosis is an essential step in the design of peer support programs that address culturally specific needs. Through one on one interviews, we hope to better understand information needs and educational preferences of individuals with inflammatory arthritis and use this information to design peer support programs that are accessible to this growing segment of our population.

II. Purpose and Objectives The specific objective of this study are to examine the learning preferences of individuals who have inflammatory arthritis, including thoughts about peer support, to identify informational needs and educational preferences related to managing arthritis and to explore how learning needs change over time or duration of the disease.

III. Methodology To explore these objectives, the perspectives of individuals with arthritis will be examined using a qualitative approach. One on one semi-structured interviews will be utilized for this component of the study.

Semi-structured Interviews Study Design Semi-structured interviews will be conducted with individuals with inflammatory arthritis acting as key informants. An interview guide (Appendix A) was developed for the purpose of this study based on a literature review of cultural needs in patient education for arthritis, previous studies of peer support needs in arthritis patients and discussion with colleagues. The interviewer will ask the same specific questions for each interview. The order of the questions may be altered and probes incorporated to obtain more information. Probes, or prompts, are questions that are not included in the interview guide, but will allow participants to elaborate on their responses and provide further discussion. Probes will be posed in a neutral manner. Depending on the data that emerges, additional questions can be added to the interview guide to obtain further information in subsequent interviews.

Data collection will continue until interviews are conducted with all key informants. There will be approximately 10-15 interviews. The interviews are anticipated to last approximately one hour each, and will be conducted by a second year medical student who is a co-investigator on this study.

Subjects

Individuals will be identified for participation in this study based on the following inclusion criteria:

* Participants must have a diagnosis of inflammatory arthritis from a physician;
* Participants must be aged 18 years or older;
* Participants must be able to participate in a 1 hour interview;
* Participants are English-speaking
* Participants are immigrants to Canada

Recruitment and Consent Process The individuals will be identified through a cohort of patients with inflammatory arthritis at a rheumatology clinic at Sunnybrook Health Sciences Centre The Principal Investigator will identify and screen potential research participants from her inflammatory arthritis patient population according to the eligibility criteria for the study and will initiate the informed consent process. The Principal Investigator will introduce the project and review the information letter for the study with each eligible patient to ensure that the potential participant understands the study and what he/she is being asked to do and to answer any questions that the potential participant may have about the study (Appendix B). The PI will obtain verbal consent for the medical student co-investigator to contact the potential research participant. When an individual has agreed to meet with the medical student co-investigator, his/her name will be forwarded to the Office Manager at the clinic. The Office Manager will contact the individual and schedule an interview at the PI's rheumatology clinic office with the medical student co-investigator assigned to the project. A confirmation letter (Appendix C) with time and location of the interview will be mailed to the participant by the Office Manager. The day before the interview is scheduled to take place the medical student will telephone the individual to remind him/her of the time and location of the interview (Appendix D). At the beginning of the interview, prior to asking any questions, the medical student will review the consent form (Appendix E) with each potential research participant to ensure that he/she understands the study and what he/she is being asked to do and answer any further questions the person may have. Once written consent is obtained, a copy will be provided to the participant.

Interviews will be conducted face-to-face. These interviews will take place at a time that is convenient for each participant in a private room at Sunnybrook Health Sciences Centre. Interviews will be tape recorded using a digital tape recorder. Transcription of each interview may occur in whole or in part. The medical student will take written notes before, during and after the interviews. These will include the student's thoughts on the interview itself, a description of any nonverbal communication by the participants, and any conversations that may not be audio-taped before or after the interviews. Personal or professional relationships between the interviewer and the participants are not anticipated.

IV. Data Analysis Interview data will be analysed using a constant comparative method of analysis. Interview data will be categorized into themes and analysed by the medical student who conducted the interviews. The transcripts will also be coded by the study coordinator and/or a second medical student, who will assist with this analysis. A preliminary coding scheme will be developed by this team, and they will first code the interview separately using this coding scheme and then meet to compare and contrast the codes. The initial interview guide may be modified with each subsequent interview to include new themes or probes that emerge in the interviews. Codes will be added to the coding scheme as new concepts are identified as the interviews progress.

V. Risks and Benefits There is a potential risk of emotional distress in patients who are asked about there illness. Should this occur, the study team will work to provide resources for support. Participants may withdraw from the study at any time without any negative consequences. Indirect benefits may be experienced due to improvement in peer support networks for arthritis patients and gained knowledge in how culture influences peer support needs of patients with arthritis.

VI. Privacy and Confidentiality Only the medical student, the research staff and the Principal Investigator involved in the study will know the identity of the key informants. No identifying information will be used on any data collections forms. For all other forms, participants will be assigned a unique identifying number. The list of names, addresses and phone numbers will be kept in a password protected computer file on a secure server in a locked research room and will only be accessed by the Principal Investigator, research staff and medical student working on the study. All information obtained during the study will be held in strict confidence. No names or identifying information will be used in any publications or presentations. No information identifying participants will be transferred outside the researchers in this study or this hospital. All of the digital files of recorded interviews will be stored as a password protected computer file on a secure server in a locked research room and deleted 25 years following completion of the study.

VII. Compensation No monetary remuneration will be provided.

VII. Communication of Results Results from this study will be communicated to an academic and health professional audience at the University of Toronto through a Determinants of Community Health (DOCH) II written report and presentation.

IX. Team Principal Investigator Mary J. Bell

Co-Investigators Joyce Nyhof-Young Lopamudra Das Romy Cho Christopher Tran Phedias Diamandis Paula Veinot

Research Assistant Gaya Embuldeniya

Study Coordinator Paula Veinot

ELIGIBILITY:
Inclusion Criteria:

Patients for one-on-one interviews:

1. Have a diagnosis of IA from a physician
2. Able to participate in a 1 hour interview
3. 18 years of age or older
4. English-speaking
5. Immigrants to Canada.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with inflammatory arthritis
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
learning needs (Informational needs and educational preferences) | o months

CONTACTS AND LOCATIONS:
Overall Officials: Mary J Bell, MD, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] References 1. Badley EM. Emerging issues. In: Arthritis and Related Conditions in Ontario: ICES Research Atlas. 2nd ed. Toronto: Institute for Clinical Evaluative Sciences; 2004. 2. Badley EM, Rasooly I, Webster GK. Relative importance of musculoskeletal disorders as a cause of chronic health problems, disability and health care utilization: Findings from the 1990 ontario health survey. Journal of Rheumatology. 1994;3(21):505-14. 3. Badley EM, Webster GK, Rasooly I. The impact of musculoskeletal disorders in the population: Are they aches and pains? findings from the 1990 ontario health survey. Journal of Rheumatology. 1995;4(22):733-9. 4. Bell M. Peer to peer mentoring program: Summary of proposed research. In press 2008. 5. Superio-Cabuslay E, Ward MM, Lorig K. Patient education interventions in osteoarthritis and rheumatoid arthritis: A meta-analytic comparison with nonsteroidal anti-inflammatory drug treatment. Arthritis Care and Research. 1996;9:292-301. 6. Health Canada. Arthritis in canada. an ongoing challenge. Ottawa: Health Canada; 2003. 7. Dennis C. Peer support within a health care context: A concept analysis. International Journal of Nursing Studies. 2003;40:321-32. 8. Osborne RH, Jordan JE, Rogers A. A critical look at the role of self-management for people with arthritis and other chronic diseases. Nature Clinical Practice Rheumatology. 2008;4:224-5. 9. Jordan JM, Lawrence R, Kingston R, Fraser P, Karlson E, Lorig K. Ethnic health disparities in arthritis and musculoskeletal diseases. report of a scientific conference. Arthritis & Rheumatology. 2002;46(9):2280-6.